CLINICAL TRIAL: NCT01962623
Title: Interpersonal Psychotherapy for Youth With Severe Mood Dysregulation- Randomized Trial
Brief Title: Interpersonal Psychotherapy for Youth With Severe Mood Dysregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Leslie Miller, M.D., Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00083893; K23MH090246 (NIH)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Severe Mood Dysregulation
Keywords: Severe Mood Dysregulation; Mood Disorders; Irritability; Disruptive Mood Dysregulation Disorder; Interpersonal Psychotherapy
MeSH Terms: conditions — Mood Disorders | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): Participants who are not randomly assigned to the IPT-MBD group will continue with treatment at usual, which is considered routine care.
  Interventions: Other: IPT-MBD
- IPT-MBD (Other): Weekly Interpersonal Therapy for SMD/DMDD (IPT-MBD) sessions, which emphasizes building skills in managing relationships, helping with problem solving, strengthening communication skills and other skills.
  Interventions: Other: IPT-MBD

INTERVENTIONS:
Other: IPT-MBD — IPT-MBD is a modified form of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A), which emphasizes building skills in managing relationships, helping with problem solving, and strengthening communication skills.
  Other Names: IPT for Mood and Behavior Dysregulation

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of utilizing an adapted form (i.e. IPT-MBD) of a psychosocial intervention, Interpersonal Psychotherapy for Depressed Adolescents, for youth with severe mood dysregulation (SMD) or disruptive mood dysregulation disorder (DMDD).

The investigators hypothesize that retention rates will be >80%, satisfaction scores will average 6 (high) on a 7 point satisfaction scale, and that youth who receive the IPT intervention will have overall improvement in SMD/DMDD symptoms.

DETAILED DESCRIPTION:
This research is being done to learn more about how to help teenagers with a sad or angry mood, and emotional responses out of proportion to what would be expected in a situation. Together these symptoms are called Severe Mood Dysregulation (SMD), a research diagnosis, or disruptive mood dysregulation disorder (DMDD), a newer clinical diagnosis. Currently, there is no standard treatment for teens that have SMD/DMDD. These teens usually receive medication and some type of talk therapy. This research is being done to compare two types of talk therapy to see which is most effective in helping teens with SMD/DMDD. Investigators will compare treatment as usual (TAU) with Interpersonal Psychotherapy for Youth with Mood and Behavior Dysregulation (IPT-MBD). Investigators do not know if TAU and IPT-MBD work just as well, or if one is better than the other. When this study is over, investigators hope there will be a better idea of how to study treatments for teens with SMD/DMDD.

For those participants who receive IPT-MBD, are prescribed an antipsychotic, and have significant improvement in symptoms, investigators will gradually taper the antipsychotic dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 12 to 17 years, who meet criteria for severe mood dysregulation (SMD) as defined by NIMH criteria or for disruptive mood dysregulation disorder (DMDD).
* Subject has an estimated IQ >70 on the Kaufman Brief Intelligence Test (KBIT-
* Subjects will have continuously resided with a legal guardian who has known the adolescent well for at least one year before study entry and is legally able to sign the consent form.
* Children's Global Assessment Scale (CGAS) ≤ 60
* CGI-S (SMD) ≥ 4
* Participant and guardian must agree to have therapy sessions audiotaped for training purposes.

Exclusion Criteria:

* Subject poses a significant risk for dangerousness to self or others. Risk will be determined by clinical history, clinical diagnostic interview and KSADS-PL interview of parent and patient by clinician.
* Subject suffers from a concomitant medical or psychiatric comorbidity that makes this study protocol inadvisable (either the treatment is contraindicated or the disorder is not the primary focus of treatment).
* Subject meets DSM-IV criteria for current alcohol or substance dependence or current use (defined as the past 4 weeks).
* Primary caretaker does not speak English or is not capable of completing study measures.
* Pregnant females.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Retention rate | 24 weeks
  To describe/assess feasibility of IPT-MBD, investigators will look at ease of recruitment and retention rate goal of at least 80%. Investigators will collect data on the number of subjects recruited, enrolled, and who followed the protocol for 24 weeks. Investigators will comment on adherence to the overall study, as well as to specific treatment visits.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale for SMD/DMDD (CGI-SMD/DMDD) | 24 weeks
  Investigators will utilize the Clinical Global Impressions Scale for Global Improvement (CGI-I) and Severity of Illness (CGI-S) to measure improvement in SMD/DMDD symptoms and to assess the effectiveness of IPT-MBD on the severity of SMD/DMDD symptoms in youth with SMD/DMDD.
Satisfaction | 24 weeks
  To assess the feasibility and acceptability of a 24-week psychosocial treatment intervention for youth with SMD/DMDD, investigators will compare satisfaction questionnaires between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Miller, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Medical Center, Baltimore, Maryland, United States